CLINICAL TRIAL: NCT01622478
Title: Validity of Sentinel Lymphnode Biopsy After Neoadjuvant Chemotherapy in Breast Cancer Patients With Radiologically Positive Axillary Lymph Nodes
Brief Title: Validity of Sentinel Lymphnode Biopsy After Neoadjuvant Chemotherapy Cancer Patients With Radiologically Positive Axillary Lymph Nodes
Acronym: VSNBNAC
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Gwe Ahn, Research Fellow, Breast Cancer Center, Gangnam Severance Hospital
Other Study IDs: GNSBCC001
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node biopsy; neoadjuvant chemotherapy; breast cancer; locally advanced breast cancer; positive axillary lymph node; negative conversion
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy; Neoadjuvant Therapy; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clinically node-positive patients before NAC: Patients with clinically positive lymph node receiving neoadjuvant chemotherapy
  1. Clinically negative-node after NAC
  2. Clinically positive-node after NAC
  Interventions: Procedure: Sentinel lymph node biopsy; Drug: Neoadjuvant chemotherapy; Procedure: complete axillary lymph node dissection; Procedure: positron emission tomography and ultrasonogram

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy — Sentinel lymph node biopsy after neoadjuvant chemotherapy for the patients with clinically positive-nodes at presentation
Drug: Neoadjuvant chemotherapy — Neoadjuvant chemotherapy for breast cancer patients with clinically positive-node at initial diagnosis
Procedure: complete axillary lymph node dissection — Complete axillary lymph node dissection after sentinel node biopsy for estimation of false-negative rate of sentinel node biopsy
Procedure: positron emission tomography and ultrasonogram — Routine evaluation of axillary nodal status using 18-fluorodeoxyglucose positron emission tomography and ultrasonogram before and after chemotherapy

SUMMARY:
Sentinel lymph node biopsy (SLNB) after neoadjuvant chemotherapy (NAC) is currently debatable. It is possible that the tumor response to chemotherapy may alter the lymphatic drainage thus causing lower SLN identification rate and higher false negative rate. Further, the response of NAC can be different in each lymph nodes. It is doubtful whether SLNB can accurately predict axillary lymph node (ALN) status after NAC. The aim of this study to determine the identification rate, the false-negative rate, and the accuracy of SLNB after NAC for node positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced breast cancer patients with node-positive proved in preoperative imaging study
* ECOG status 0-1

Exclusion Criteria:

* No previous cancer history
* No previous chemotherapy history

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Advanced breast cancer patients with node-positive proved in preoperative imaging study
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, Seoul, South Korea